CLINICAL TRIAL: NCT05888402
Title: The Efficacy and Safety of Induction Chemotherapy and Toripalimab Followed by Chemoradiotherapy for Large-volume (Bulky) Local Advanced Non-small Cell Lung Cancer
Brief Title: Induction Chemotherapy and Toripalimab Followed by Chemoradiotherapy for Large-volume Local Advanced NSCLC
Acronym: InTRist
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: InTRist
Record Dates: First submitted 2023-03-18; First posted 2023-06-05 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2022-11

CONDITIONS: Local Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction Toripalimab and chemotherapy followed by concurrent chemoradiotherapy (Experimental): Participants will receive 2 cycles of induction therapy of platinum-based chemotherapy combined with Toripalimab, followed by platinum-based concurrent chemoradiation. Then participants will receive Toripalimab consolidation therapy after chemoradiotherapy with maximum 1 years or until disease progression or intolerable toxicity.
  Interventions: Drug: Toripalimab; Radiation: Concurrent chemoradiation therapy and consolidation immunotherapy
- Induction chemotherapy followed by concurrent chemoradiotherapy (Active Comparator): Participants will receive 2 cycles of induction platinum-based chemotherapy, followed by platinum-based concurrent chemoradiation. Then participants will receive Toripalimab consolidation therapy after chemoradiotherapy with maximum 1 years or until disease progression or intolerable toxicity.
  Interventions: Radiation: Concurrent chemoradiation therapy and consolidation immunotherapy

INTERVENTIONS:
Drug: Toripalimab — Two cycles of induction Toripalimab (240mg every 3 weeks) plus platinum-based doublet chemotherapy as induction chemoimmunotherapy.
  Other Names: Tuo Yi
  Arms: Induction Toripalimab and chemotherapy followed by concurrent chemoradiotherapy
Radiation: Concurrent chemoradiation therapy and consolidation immunotherapy — Thoracic radiation therapy (54-66Gy/25-33F/5-7week), concurrently with platinum-based doublet chemotherapy, followed by consolidation Toripalimab (240mg every 3 weeks) as consolidation immunotherapy for up to 12 months.
  Other Names: The PACIFIC regimen

SUMMARY:
This study is a Phase II study to evaluate the clinical efficacy and safety of Toripalimab combined with chemoradiotherapy for large-volume local advanced non-small cell lung cancer

DETAILED DESCRIPTION:
This study is a Phase II study to evaluate the clinical efficacy and safety of two cycles of induction Toripalimab plus chemotherapy followed by definitive chemoradiotherapy and consolidation Toripalimab therapy for large-volume, unresectable, locally advanced stage II-III non-small cell lung cancer ("large volume" is defined as primary tumor ≥5 cm in greatest dimension or metastatic lymph nodes ≥2 cm in shortest diameter).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years; ECOG score 0-2.
2. Histologically or cytologically confirmed non-small cell lung cancer (NSCLC).
3. Unresectable Stage II-III NSCLC (according to AJCC 8th edition) with maximum tumor diameter T ≥ 5 cm in the primary tumor or minimum diameter N ≥ 2 cm in mediastinal metastatic lymph nodes.
4. No other previous anti-tumor history, at least 3 months of expected survival.
5. No serious medical diseases and dysfunction of major organs, such as blood routine, liver, kidney, heart and lung function.

Exclusion Criteria:

1. Pathologic type was adenocarcinoma with EGFR gene mutation or ALK gene rearrangement.
2. Patients with other active malignancies within 5 years or at the same time.
3. Active or previously documented autoimmune or inflammatory diseases (including inflammatory bowel disease, diverticulitis [except diverticular disease], systemic lupus erythematosus, Sarcoidosis syndrome, Wegener' s syndrome).
4. History of allogeneic organ transplantation.
5. History of active primary immunodeficiency.
6. Patients with uncontrolled concurrent diseases, including but not limited to persistent or active infection (including tuberculosis, hepatitis B, hepatitis C, human immunodeficiency virus, etc.), symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled arrhythmia, active interstitial lung disease, severe chronic gastrointestinal disease with diarrhea or mental illness.
7. Women of child-bearing potential who are pregnant or breastfeeding.
8. Allergic to research drug ingredients.
9. Ongoing or prior use of immunosuppressive agents within 14 days prior to first dose
10. The investigator judged other situations not suitable for inclusion in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of recruitment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Defined as the time from date of recruitment until the date of first documented progression or date of death from any cause, whichever came first.

SECONDARY OUTCOMES:
Overall survival (OS） | From recruitment to the date of any documented death due to any cause, assessed up to 36 months.
  Defined as the time from recruitment to the date of any documented death due to any cause.
Adverse Event | AEs and SAEs must be collected from the time that the main study informed consent is obtained to 28 days after discontinuation of study drug, up to 36 months.
  The incidence of adverse events (AEs) and serious adverse events (SAEs), evaluated by CTCAE 5.0. Appropriate description of AEs and laboratory data/vital signs will be produced. Number of patients who had at least one adverse event will be calculated.
Objective Tumour Response (ORR) | Tumor assessment using RECIST will be performed at baseline then every 42 days (6 weeks) ± 7 days (1 week) from recruitment until objective progression or death from any cause, assessed up to 36 months.
  The objective tumour response (ORR) will be calculated as the number of patients with CR or PR per RECIST Criteria. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Disease control rate（DCR） | Tumour assessment using RECIST will be performed at baseline then every 42 days (6 weeks) ± 7 days (1 week) from randomisation until objective progression or death from any cause, assessed up to 36 months.
  DCR will be calculated as the number of patients with CR, PR or sustained SD≥6 weeks per RECIST Criteria. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Bi, MD, Principal Investigator — Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Deng L, Wang J, Zhang T, Wang W, Wang X, Liu W, Wu Y, Lv J, Feng Q, Zhou Z, Wang J, Wang L, Wang Z, Bi N. Induction PD-1 inhibitor toripalimab plus chemotherapy followed by concurrent chemoradiotherapy and consolidation toripalimab for bulky locally advanced non-small-cell lung cancer: protocol for a randomized phase II trial (InTRist study). Front Immunol. 2024 Jan 15;14:1341584. doi: 10.3389/fimmu.2023.1341584. eCollection 2023. PMID 38288117